CLINICAL TRIAL: NCT03388645
Title: Challenge Infection of Healthy Adult Volunteers With RSV A2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 180039; 18-I-0039
Record Dates: First submitted 2017-12-30; First posted 2018-01-03 (Actual); Results first posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2019-12-06

CONDITIONS: Upper Respiratory Tract Infections
Keywords: RSV Shedding; Immune Responses; Neutralizing Antibody Titer; Upper Respiratory Tract Infection
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Low Dose 10^6.3 PFU of RSV A2 (Experimental): Single intranasal dose of 10^6.3 plaque forming units (PFU) of respiratory syncytial virus A2 (RSV A2) using a nasal atomizer on Day 0
  Interventions: Biological: 10^6.3 PFU of RSV A2
- High Dose 10^7 PFU of RSV A2 (Experimental): Single intranasal dose of 10^7 plaque forming units (PFU) of respiratory syncytial virus A2 (RSV A2) using a nasal atomizer on Day 0
  Interventions: Biological: 10^7 PFU of RSV A2

INTERVENTIONS:
Biological: 10^6.3 PFU of RSV A2 — Each adult volunteer will receive a single intranasal inoculation of 10^6.3 PFU of RSV A2 administered with a nasal atomizer with subsequent sampling of nasal fluids and blood draws.
  Arms: Low Dose 10^6.3 PFU of RSV A2
Biological: 10^7 PFU of RSV A2 — Each adult volunteer will receive a single intranasal inoculation of 10^7 PFU of RSV A2 administered with a nasal atomizer with subsequent sampling of nasal fluids and blood draws.
  Arms: High Dose 10^7 PFU of RSV A2

SUMMARY:
Background:

One of the main causes of respiratory infections in children and adults is RSV. This stands for respiratory syncytial virus. Healthy adults usually get a cold when they get an infection with RSV. They generally recover without any problems. But some infections can be life-threatening. Researchers want to study RSV infection in a safe, controlled setting in healthy adults to help develop new treatments.

Objective:

To test the safety of a high dose of RSV A2 by spraying the virus into the nose, and studying how the body responds.

Eligibility:

Healthy adults ages 18-50

Design:

Participants will be screened during 2 screening visits with:

* Medical interview
* Physical exam
* Blood and nasal samples
* Chest X-ray (chest radiograph)
* Participants will have a heart test. Sticky patches on the body will detect heart electrical activity.
* Pulmonary function test (PFT). They will blow into a machine to measure airflow.
* Urine tests for pregnancy or drug use.

Participants will be admitted to the hospital before they get RSV A2.

Participants will get a single dose of RSV A2 as two sprays, one into each nostril.

Participants will stay in the hospital under isolation for as long as it takes the body to clear RSV A2 from nasal fluids. This can take as long as 14 days or more.

Participants cannot take any cold medicine to try to feel better.

Every day, participants will:

* Answer questions about their symptoms
* Have nasal washes and/or nasal swabs collected
* Have a physical exam

Participants will have blood drawn most days.

After discharge, participants will keep a health diary.

Participants will have 2 follow-up visits at 1 month and 2 months after receiving the RSV A2 dose. A history and physical examination, a blood draw, and nasal wash and swab will be performed.

DETAILED DESCRIPTION:
Respiratory syncytial virus (RSV) is the leading cause of pediatric lower respiratory tract infection. RSV also causes lower respiratory tract disease in the elderly and life-threatening disease in immunocompromised hosts. An RSV monoclonal antibody (palivizumab) is currently available for passive immunoprophylaxis in high-risk infants. Vaccines and antiviral agents are under development for the treatment and prevention of RSV, but none are licensed. The ability to challenge healthy volunteers with RSV could rapidly facilitate efficacy studies of future antivirals and vaccines. In addition, challenge studies would provide critical information on viral pathogenesis, including types of cells infected, mucosal and systemic immune response, and alterations in respiratory microbiota. Clinical trial material for human challenge studies has been prepared from live recombinant (complementary DNA-derived) RSV of subgroup A (RSV A2).

This study will be a phase 1 study in healthy adult male and non-pregnant female subjects 18 years to 50 years of age. The main purpose of the trial is to define the safety profile, determine the frequency of RSV shedding in nasal wash, estimate RSV illness rates, and study immune responses in subjects given 1 dose of 10^7 PFU of RSV A2 challenge virus using a nasal atomizer. If RSV A2 is found to be sufficiently infectious in adults, then it may be used as a challenge virus in future studies evaluating antivirals or the protective efficacy of RSV vaccines, or in studies of the immunopathogenesis of RSV infection.

Subjects will be admitted to the NIH Clinical Center and receive a single intranasal dose of 10^6.3 PFU or 107 PFU of RSV A2. Subjects will remain at the Clinical Center for approximately 9-14 days after challenge infection undergoing sequential clinical evaluations. Research specimens, nasal washes and blood, will be collected for various research assays. Subjects will be discharged when their daily nasal wash RSV result is negative for two days in a row, and they do not have any signs or symptoms suggestive of possible RSV-associated lower respiratory tract disease. Subjects will return for follow-up evaluation 28 and 56 days after viral challenge.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Age 18-50 years inclusive.
  2. General good health, without significant medical illness, physical exam findings, or significant laboratory abnormalities as determined by the investigator.
  3. Willingness to stay confined to the inpatient unit for required study duration.
  4. Willingness to have samples stored for future research.
  5. Subjects must be of non-childbearing potential (e.g., surgically sterilized (bilateral oophorectomy, bilateral tubal ligation, hysterectomy) or, if of child-bearing potential and sexually active with a partner who can get them pregnant, must have in place an effective method of contraception for at least 30 days prior to administration of the challenge virus and until 30 days after challenge virus

     administration:
     * intrauterine device (IUD) or equivalent
     * hormonal contraceptives (e.g., consistent, continuous use of contraceptive pill, patch, ring, implant, or injection)

       ---if participant uses contraceptive pill, patch, or ring, they must also use a barrier method at the time of potentially reproductive sexual activity (e.g., (male/female condom, cap, or diaphragm) plus spermicide)
     * be in a monogamous relationship with a partner who has undergone a vasectomy at least 180 days prior to first dose of study agent
  6. A plaque reduction RSV neutralization titer < 8.0 log(2).

EXCLUSION CRITERIA:

1. Subject who was previously challenged with RSV A2.
2. Female subject who is pregnant or lactating OR planning to become pregnant from 30 days prior to inoculation through 30 days after inoculation.
3. Presence of self-reported or medically documented significant medical condition(s) including but not limited to:

   -Respiratory disease (e.g., chronic obstructive pulmonary disease, emphysema, rhinitis, sinusitis) in adulthood, and additionally:

   --A history of asthma within the past 5 years, or a current diagnosis of asthma or reactive airway disease associated with

   exercise, seasonal hay fever or allergic rhinitis

   --Presence of any febrile illness or symptoms suggestive of a respiratory infection within 2 weeks prior to inoculation.
   * Any significant abnormality of the nose or nasopharynx, including recurrent epistaxis within 90 days prior to viral inoculation or nasal or sinus surgery within 180 days prior to viral inoculation.
   * Chronic cardiovascular disease (e.g., congestive heart failure, cardiomyopathy, ischemic heart disease).
   * Chronic neurological or neurodevelopmental conditions (e.g., cerebral palsy, epilepsy, stroke, seizures).
   * Ongoing malignancy.
   * Chronic medical condition requiring close medical follow-up or hospitalization during the past 5 years (e.g., diabetes mellitus, renal dysfunction, hemoglobinopathy, autoimmune disease).
   * An immunodeficiency.
4. Use of systemic corticosteroids exceeding 10 mg/day of prednisone equivalent and nasal steroid preparations or immunosuppressive drugs within 30 days before inoculation and within 60 days after. Low dose topical steroid preparations used for a discrete period of time are permitted.
5. Inhaled bronchodilator or inhaled steroid use within the last 360 days or use after upper respiratory tract infections.
6. Behavioral or cognitive impairment or psychiatric disease that in the opinion of the investigator affects the ability of the subject to understand and cooperate with the study protocol.
7. Complete blood count (CBC), aspartate aminotransferase (AST), alanine aminotransferase (ALT), creatinine values or other screening labs or tests (e.g. electrocardiogram (EKG), chest x-ray (CXR)) are outside of the NIH Department of Laboratory Medicine normal reference range and deemed clinically significant by the PI.
8. Positive FDA-approved HIV test obtained during screening procedures.
9. Positive serology for hepatitis C virus obtained during screening period.
10. Presence of hepatitis B surface antigen obtained during screening period.
11. A smoker of tobacco products or a routine marijuana smoker currently or in the past year.
12. Current alcohol abuse or addiction.
13. Current illicit drug abuse or addiction.
14. Receipt of a licensed vaccine within 30 days prior to RSV A2 inoculation and planned vaccination within 60 days after inoculation..
15. Receipt of blood or blood-derived products (including immunoglobulin) within 180 days prior to viral inoculation. Receipt of packed red blood cells given for an emergent indication in an otherwise healthy person, and not required as ongoing treatment, is not exclusionary.
16. Receipt of an investigational agent or vaccine within 90 days prior to scheduled RSV A2 inoculation and planned receipt within 60 days after inoculation.
17. A body mass index (BMI) less than or equal to 18.5 or greater than or equal to 37.0.
18. A medical, occupational, or family problem that would preclude the participant from complying with all study requirements.
19. Shares household, works closely with, or has routine contact with a child (children) < 5 years of age or with immunocompromised individual(s), adult(s) with significant cardiopulmonary disease or asthma, institutionalized persons or persons with functional disability, or any other individual that, in the judgment of the PI, might be at increased risk for complications if exposed to RSV.
20. Deprived of freedom by an administrative or court order or in an emergency setting.
21. Any condition that in the opinion of the PI would jeopardize the safety or rights of a person participating in the trial or would render the person unable to comply with the protocol.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lesia K Dropulic, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] DeVincenzo JP, Whitley RJ, Mackman RL, Scaglioni-Weinlich C, Harrison L, Farrell E, McBride S, Lambkin-Williams R, Jordan R, Xin Y, Ramanathan S, O'Riordan T, Lewis SA, Li X, Toback SL, Lin SL, Chien JW. Oral GS-5806 activity in a respiratory syncytial virus challenge study. N Engl J Med. 2014 Aug 21;371(8):711-22. doi: 10.1056/NEJMoa1401184. PMID 25140957
- [Background] Hall CB, Long CE, Schnabel KC. Respiratory syncytial virus infections in previously healthy working adults. Clin Infect Dis. 2001 Sep 15;33(6):792-6. doi: 10.1086/322657. Epub 2001 Aug 21. PMID 11512084
- [Background] Lee FE, Walsh EE, Falsey AR, Betts RF, Treanor JJ. Experimental infection of humans with A2 respiratory syncytial virus. Antiviral Res. 2004 Sep;63(3):191-6. doi: 10.1016/j.antiviral.2004.04.005. PMID 15451187
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2018-I-0039.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 19 subjects were recruited; 7 were not dosed because they were either ineligible or did not start the study.
Period: Low Dose RSV A2
Arm/Group | Low Dose 10^6.3 PFU of RSV A2 | High Dose 10^7 PFU of RSV A2
Started | 4 | 0
Completed | 4 | 0
Not Completed | 0 | 0
Period: High Dose RSV A2
Arm/Group | Low Dose 10^6.3 PFU of RSV A2 | High Dose 10^7 PFU of RSV A2
Started | 0 | 8
Completed | 0 | 7
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose 10^6.3 PFU of RSV A2 | High Dose 10^7 PFU of RSV A2 | Total
Number analyzed (Participants) | 4 | 8 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 8 | 12
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 3 | 4 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 2 | 7 | 9
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 3 | 5 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Participants With Detectable RSV Shedding in Nasopharyngeal Wash
Description: Participants who had shedding of RSV as assessed by detection of RSV A2 in nasal wash by FilmArray multiplex polymerase chain reaction (PCR), by reverse transcriptase (RT)-quantitative PCR, or by quantitative viral culture.
Time Frame: Daily from study Day 2 through day 10 after challenge with RSV A2
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose 10^6.3 PFU of RSV A2 | High Dose 10^7 PFU of RSV A2
Number analyzed (Participants) | 4 | 8
Participants | 2 | 4

2. Primary Outcome: Participants With Related, Expected Adverse Events After Challenge
Description: Participants who had one or more episodes of related, expected adverse events. Participants were evaluated for grades 1 to 3 adverse events. Only grade 1 adverse events were experienced.
Time Frame: Safety assessed continuously during the inpatient phase and at Day 28 and 56 during the outpatient phase of the study
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose 10^6.3 PFU of RSV A2 | High Dose 10^7 PFU of RSV A2
Number analyzed (Participants) | 4 | 8
Participants
  Nasal congestion or rhinorrhea | 3 | 2
  Sore throat | 2 | 4
  Cough | 0 | 3
  Headache | 2 | 0
  Sinus congestion or pain | 1 | 1
  Fever 38°C to 39.4°C | 0 | 0
  Ear Pain | 0 | 0

3. Primary Outcome: Participants With Unrelated Expected Adverse Events After Challenge
Description: Participants who had one or more episodes of unrelated, expected adverse events. Participants were evaluated for grades 1 to 3 adverse events. Only grade 1 adverse events were experienced.
Time Frame: Safety assessed continuously during the inpatient phase and at Day 28 and 56 during the outpatient phase of the study
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose 10^6.3 PFU of RSV A2 | High Dose 10^7 PFU of RSV A2
Number analyzed (Participants) | 4 | 8
Participants
  Nasal congestion or rhinorrhea | 1 | 0
  Headache | 1 | 1
  Cough | 1 | 1
  Sinus congestion or pain | 0 | 1

4. Primary Outcome: Participants With Related, Unexpected Adverse Events After Challenge
Description: Participants who had one or more episodes of related, unexpected adverse events. Related, unexpected adverse events are those that are not expected but are related to RSV A2 or of grade 4 severity and related to RSV A2. Only grade 1 adverse events were experienced.
Time Frame: Safety assessed continuously during the inpatient phase and at Day 28 and 56 during the outpatient phase of the study
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose 10^6.3 PFU of RSV A2 | High Dose 10^7 PFU of RSV A2
Number analyzed (Participants) | 4 | 8
Participants
  Alanine aminotransferase | 1 | 0
  Anxiety | 1 | 0
  Bradycardia | 2 | 0
  Chills | 0 | 1
  Fatigue | 0 | 1
  General discomfort | 0 | 1
  Postnasal drip | 1 | 0
  Respiratory rate | 1 | 0
  Smell alteration | 0 | 1
  Sneezing | 0 | 2
  Taste alteration | 0 | 1
  Throat irritation | 0 | 4
  Watering eyes | 1 | 0

5. Primary Outcome: Participants With Unrelated, Unexpected Adverse Events After Challenge
Description: Participants who had one or more episodes of unrelated, unexpected adverse events. Unrelated, unexpected adverse events are those that are not expected and are not related to RSV A2.
Time Frame: Safety assessed continuously during the inpatient phase and at Day 28 and 56 during the outpatient phase of the study
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose 10^6.3 PFU of RSV A2 | High Dose 10^7 PFU of RSV A2
Number analyzed (Participants) | 4 | 8
Participants
  Abdominal pain | 0 | 1
  Bradycardia | 1 | 2
  Bruising aminotransferase | 1 | 0
  Cognitive disturbance | 1 | 0
  Hemoglobin decreased | 1 | 5
  Irritability | 1 | 0
  Laceration | 1 | 0
  Light headedness | 0 | 2
  Low back pain | 1 | 0
  Muscle soreness | 0 | 1
  Nausea | 1 | 0
  Neck pain | 1 | 0
  Night sweats | 1 | 0
  Pain | 1 | 0
  Potassium decreased | 0 | 1
  Syncope | 0 | 1
  Tiredness | 0 | 1

6. Secondary Outcome: Participants With Mild to Moderate Upper Respiratory Illness
Description: Participants who experienced mild to moderate upper respiratory illness in healthy volunteers challenged with RSV A2. All RSV illness qualified as mild illness.
Time Frame: Daily from study Day 2 through day 10 after RSV challenge
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose 10^6.3 PFU of RSV A2 | High Dose 10^7 PFU of RSV A2
Number analyzed (Participants) | 4 | 8
Participants | 2 | 1

ADVERSE EVENTS:
Time Frame: 56 days
Arm/Group | Low Dose 10^6.3 PFU of RSV A2 | High Dose 10^7 PFU of RSV A2
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/8
Other Adverse Events (participants affected / at risk) | 4/4 | 7/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose 10^6.3 PFU of RSV A2 (N=4) | High Dose 10^7 PFU of RSV A2 (N=8)
Bradycardia (Cardiac disorders) | 2 | 2
Lacrimation increased (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Chills (General disorders) | 0 | 1
Discomfort (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 2
Pain (General disorders) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Blood potassium decreased (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 1 | 4
Respiratory rate (Investigations) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 2
Headache (Nervous system disorders) | 3 | 1
Parosmia (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Taste disorder (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Irritability (Psychiatric disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-08): https://cdn.clinicaltrials.gov/large-docs/45/NCT03388645/Prot_SAP_000.pdf